CLINICAL TRIAL: NCT02553330
Title: An Open-Label (Part A) and a Double-Blind, Randomized, Placebo Controlled (Part B) Study, With an Open-Label Extension, of Ruxolitinib Phosphate Cream Applied Topically to Subjects With Alopecia Areata
Brief Title: A Study With Ruxolitinib Phosphate Cream Applied Topically to Subjects With Alopecia Areata (AA)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early based on the results of a planned interim analysis.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCB 18424-204
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Alopecia Areata
Keywords: Hair loss; alopecia areata; alopecia totalis; alopecia universalis; JAK inhibitors; topical hair growth
MeSH Terms: conditions — Alopecia Areata; Alopecia; Alopecia universalis | interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ruxolitinib Phosphate Cream (Experimental): Part A: Open-label treatment is 24 weeks, an optional open-label treatment extension is 24 weeks if eligible, and follow-up is an additional 12 weeks;
  Part B: Double-blind treatment is 24 weeks, an optional open-label treatment extension is 24 weeks if eligible, and follow-up is an additional 12 weeks.
  Interventions: Drug: Ruxolitinib Phosphate Cream
- Placebo Cream (Placebo Comparator): Part B: Double-blind treatment is 24 weeks (and/or treatment with Ruxolitinib Phosphate Cream if eligible) and follow-up is an additional 12 weeks.
  Interventions: Drug: Placebo Cream; Drug: Ruxolitinib Phosphate Cream

INTERVENTIONS:
Drug: Placebo Cream
  Arms: Placebo Cream
Drug: Ruxolitinib Phosphate Cream
  Other Names: INCB018424

SUMMARY:
A phase 2 study to find out if the drug ruxolitinib Phosphate Cream is safe and has beneficial effects in people who have alopecia areata (partial or complete hair loss) when applied to the skin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AA
* Duration and extent of current episode of AA
* Evidence of active hair loss

Exclusion Criteria:

* Evidence of diffuse, spontaneous terminal hair regrowth
* Receipt of treatment known to potentially affect the course of AA within last month

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Butler, MD, Study Director — Incyte Corporation
Locations (18):
- United States (18):
  - Birmingham, Alabama
  - Hot Springs, Arkansas
  - New Haven, Connecticut
  - Trumbull, Connecticut
  - Miami, Florida
  - Beverly, Massachusetts
  - Boston, Massachusetts
  - Clinton Township, Michigan
  - Fort Gratiot, Michigan
  - Fridley, Minnesota
  - Minneapolis, Minnesota
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Portland, Oregon
  - Austin, Texas
  - Houston, Texas
  - Katy, Texas
  - Norfolk, Virginia

REFERENCES:
- [Derived] Bayart CB, DeNiro KL, Brichta L, Craiglow BG, Sidbury R. Topical Janus kinase inhibitors for the treatment of pediatric alopecia areata. J Am Acad Dermatol. 2017 Jul;77(1):167-170. doi: 10.1016/j.jaad.2017.03.024. No abstract available. PMID 28619556

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 17 study centers in the United States.
Pre-assignment Details: Twelve participants were enrolled at 4 sites and were evaluable in the Part A treatment period; In Part B, 78 additional participants were enrolled at 17 sites.
Groups:
- Part A: Ruxolitinib Cream: Part A: Open-label treatment is 24 weeks, an optional open-label treatment extension is 24 weeks if eligible, and follow-up is an additional 12 weeks
- Part B : Placebo Cream: Part B: Double-blind treatment is 24 weeks and/or optional treatment with Ruxolitinib Phosphate Cream if eligible and follow-up is an additional 12 weeks
- Part B : Ruxolitinib Cream: Part B: Double-blind treatment is 24 weeks, an optional open-label treatment extension is 24 weeks if eligible, and follow-up is an additional 12 weeks.
Period: Overall Study
Arm/Group | Part A: Ruxolitinib Cream | Part B : Placebo Cream | Part B : Ruxolitinib Cream
Started | 12 | 39 | 39
Completed | 7 | 0 | 2
Not Completed | 5 | 39 | 37
Not completed — Study Terminated by Sponsor | 2 | 13 | 12
Not completed — Withdrawal by Subject | 3 | 19 | 21
Not completed — Other | 0 | 1 | 0
Not completed — Non compliance to study treatment | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Ruxolitinib Cream | Part B : Placebo Cream | Part B : Ruxolitinib Cream | Total
Number analyzed (Participants) | 12 | 39 | 39 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.6 (13.17) | 44.3 (15.92) | 42.4 (14.69) | 43.4 (15.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 24 | 27 | 60
  Male | 3 | 15 | 12 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 11 | 33 | 29 | 73
  Black or African American | 0 | 5 | 4 | 9
  Asian | 1 | 1 | 0 | 2
  Other | 0 | 0 | 5 | 5
  Unknown | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 5 | 9
  Not Hispanic or Latino | 11 | 36 | 33 | 80
  Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part A: Percentage of Participants Achieving a ≥ 50% Improvement in SALT50 Response in Terminal Hair (Pigmented and Nonpigmented).
Description: Percentage of subjects achieving a SALT 50 (defined as a ≥ 50% improvement from baseline in SALT). SALT score is on a percent scale where 0% is no hair loss and 100 % is total hair loss.
Time Frame: Up to Week 24
Population: Part A evaluable population in treatment period includes all subjects exposed to at least 1 dose of study drug in that period.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Ruxolitinib Cream
Number analyzed (Participants) | 12
Participants
  Week 4 | 0
  Week 8 | 0
  Week 12 | 3
  Week 18 | 4
  Week 24 | 6

2. Primary Outcome: Part B : Percentage of Participants Achieving a SALT50 Response in Terminal Hair (Pigmented and Nonpigmented)
Description: as for outcome 1
Time Frame: Week 24
Population: Intent to Treat population in the Part B treatment period i.e all participants who are randomized
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Ruxolitinib Cream: Part B: Double-blind treatment is 24 weeks, an optional open-label treatment extension is 24 weeks if eligible, and follow-up is an additional 12 weeks.
Arm/Group | Part B : Placebo Cream | Part B: Ruxolitinib Cream
Number analyzed (Participants) | 39 | 39
Participants | 5 | 5

3. Secondary Outcome: Part A : Percentage of Participants With 50% to 100% Scalp Involvement at Baseline Achieving a SALT50 Response in Terminal Hair.
Description: Number of participants achieving 50% or greater improvement in their SALT score (SALT50) compared to Baseline. SALT score 0-100 with lower score indicating better health outcomes.
Time Frame: Up to Week 24
Population: The subgroup analysis was performed on subjects exposed to at least 1 dose of study drug in that period with a baseline SALT score of 50-100%.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Ruxolitinib Cream
Number analyzed (Participants) | 7
Participants
  Week 4 | 0
  Week 8 | 0
  Week 12 | 2
  Week 18 | 3
  Week 24 | 4

4. Secondary Outcome: Part B : Percentage of Participants With 50% to 100% Scalp Involvement at Baseline Achieving a SALT50 Response in Terminal Hair (Pigmented and Nonpigmented).
Description: as for outcome 3
Time Frame: Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part B : Placebo Cream | Part B : Ruxolitinib Cream
Number analyzed (Participants) | 22 | 21
Participants | 2 | 4

5. Secondary Outcome: Part A and B : Percentage of Participants Achieving a SALT90 Response in Terminal Hair.
Description: Number of participants achieving 90% or greater improvement in their SALT score (SALT90) compared to Baseline. SALT score 0-100 with lower score indicating better health outcomes.
Time Frame: Weeks 4, 8, 12, 18, and 24.
Population: Part A evaluable population in treatment period includes all subjects exposed to at least 1 dose of study drug in that period.
  Intent to Treat population in the Part B treatment period i.e all participants who are randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Ruxolitinib Cream | Part B : Placebo Cream | Part B : Ruxolitinib Cream
Number analyzed (Participants) | 12 | 39 | 39
Participants
  Week4 | 0 | 0 | 0
  Week 8 | 0 | 0 | 0
  Week 12 | 0 | 0 | 1
  Week 18 | 1 | 0 | 2
  Week 24 | 2 | 0 | 2

6. Secondary Outcome: Part B : Percentage of Subjects Whose AA Lesions Treated Since Baseline Achieved a Physician's Global Assessment of Regrowth (PGARG) Score of at Least 3
Description: Number of subjects achieving a Physician's Global Assessment (PGA) score of 3 or above at week 24 (0, no regrowth; 1, <25% of regrowth; 2, 25%-49% of regrowth; 3, 50%-74% of regrowth; 4, 75%-99% of re- growth; 5, 100% of regrowth).
Time Frame: Baseline to Week 24
Population: Intent to Treat population in the Part B treatment period i.e all participants who are randomized. Participants dropped out of study by week 24 were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B : Placebo Cream | Part B : Ruxolitinib Cream
Number analyzed (Participants) | 33 | 33
Participants | 5 | 2

7. Secondary Outcome: Part B : Percentage of Participants Achieving a SALT50 in Terminal Hair (Pigmented and Nonpigmented).
Description: as for outcome 3
Time Frame: Weeks 4, 8, 12, and 18.
Population: Intent to Treat population in the Part B treatment period i.e all participants who are randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B : Placebo Cream | Part B : Ruxolitinib Cream
Number analyzed (Participants) | 39 | 39
Participants
  Week 4 | 0 | 0
  Week 8 | 0 | 2
  Week 12 | 1 | 3
  Week 18 | 4 | 5

8. Secondary Outcome: Part B: Mean Change From Baseline in SALT Score
Description: Severity of Alopecia Tool Score (SALT) calculation is based on a scoring system. The scalp is divided into the following 4 areas: 1) Vertex: 40% (0.4) of scalp surface area, 2) Right profile of scalp: 18% (0.18) of scalp surface area, 3) Left profile of scalp: 18% (0.18) of scalp surface area, and 4) Posterior aspect of scalp: 24% (0.24) of scalp surface area. The percentage of hair loss in any of these areas is the percentage hair loss multiplied by percent surface area of the scalp in that area. The SALT score is the sum of percentage of hair loss in all the above-mentioned areas, so a lower number indicates a better outcome. The reported SALT score range is from a minimum of 0 (no hair loss) to a maximum of 100 (100% hair loss).
Time Frame: Weeks 4, 8, 12, 18, and 24.
Population: Intent to Treat population in the Part B treatment period i.e all participants who are randomized.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Part B : Placebo Cream | Part B : Ruxolitinib Cream
Number analyzed (Participants) | 39 | 39
Units on a Scale
  Change from Baseline to Week 4: number analyzed (Participants) | 36 | 38
  Change from Baseline to Week 4 | 1.02 (1.577) | 0.13 (1.534)
  Change from Baseline to Week 8: number analyzed (Participants) | 35 | 38
  Change from Baseline to Week 8 | 2.13 (2.233) | -1.11 (2.160)
  Change from Baseline to Week 12: number analyzed (Participants) | 34 | 35
  Change from Baseline to Week 12 | 1.23 (2.956) | -2.55 (2.873)
  Change from Baseline to Week 18: number analyzed (Participants) | 33 | 33
  Change from Baseline to Week 18 | -0.01 (3.550) | -4.16 (3.461)
  Change from Baseline to Week 24: number analyzed (Participants) | 33 | 33
  Change from Baseline to Week 24 | -1.68 (3.886) | -3.92 (3.794)

9. Secondary Outcome: Part A and B : Number of Treatment-emergent Adverse Events
Description: Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment
Time Frame: Up to 100 weeks
Population: All enrolled subjects who received at least 1 dose of INCB018424 or Placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Ruxolitinib Cream | Part B : Placebo Cream | Part B : Ruxolitinib Cream
Number analyzed (Participants) | 12 | 38 | 39
Participants
  Treatment Period | 9 | 28 | 23
  Extension Period: number analyzed (Participants) | 9 | 32 | 31
  Extension Period | 7 | 23 | 22

ADVERSE EVENTS:
Time Frame: Up to 100 weeks
Description: The safety population included all randomized subjects who received at least 1 dose of study drug.
Groups:
- Placebo Cream: Part B: Double-blind treatment for 24 weeks.
- Ruxolitinib Cream: Part A: Open-label treatment for 24 weeks. Part B: Double-blind treatment for 24 weeks. Placebo group from Part B had the option to crossover after the first 24 weeks of treatment period.
  Both Part A and Part B participants, if eligible, continued on to open-label extension (24 weeks) and long-term extension (48 weeks) periods.
Arm/Group | Placebo Cream | Ruxolitinib Cream
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/38 | 4/83
Other Adverse Events (participants affected / at risk) | 14/38 | 31/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cream (N=38) | Ruxolitinib Cream (N=83)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cream (N=38) | Ruxolitinib Cream (N=83)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 6 (6) | 13 (16)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 10 (11)
Sinusitis (Infections and infestations) | 1 (1) | 7 (7)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT02553330/Prot_000.pdf
  • Statistical Analysis Plan (2015-10-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT02553330/SAP_001.pdf